CLINICAL TRIAL: NCT06703307
Title: Identifying Biomarkers Related to Post-stroke Cognitive Impairment: A fNIRS Study
Brief Title: Biomarkers Related to PSCI: An fNIRS Study
Status: Recruiting | Type: Observational
Sponsor: Dingqun Bai (Other)
Responsible Party: Sponsor-Investigator, Dingqun Bai, Director of rehabilitation Medicine, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 20241121
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Cognitive Decline
Keywords: stroke; post-stroke cognitive impairment; fNIRS
MeSH Terms: conditions — Stroke; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy subjects: Healthy subjects without history of stroke or cognitive impairment.
- PSCI: Stroke patients with post-stroke cognitive impairment.
- NPSCI: Stroke patients without post-stroke cognitive impairment.

SUMMARY:
This is an fNIRS study performed to identify biomarkers related to post-stroke cognitive impairment.

DETAILED DESCRIPTION:
This was an initial screening and preliminary intervention study. Both healthy subject and stroke patients will be included in this study. Brain functional activation of each subject during the cognitive task (Stroop task, 1-back task and verbal fluency test) will be evaluated using functional near-infrared spectroscopy (fNIRS). Cognitive function related scale assessment included Mental State Examination Scale (MMSE), Montreal Cognitive Assessment (MoCA), drawing clock test (DCT), Shape trials test A.B (STT-A, STT-B), standardized digital modal test (SDMT), auditory verbal learning test-Huashan version (AVLT-H), and activity of daily living (ADL) scale will be used to evaluate the function of each patient. Biomarkers related to post-stroke cognitive impairment will be identified by by comparing differences in brain activation and brain network connectivity between patients and healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

Stroke patients:

1. Diagnosis of stroke confirmed by neuroimaging (CT or MRI)
2. 18-80 years old
3. Able to complete the cognitive task
4. Able to follow instructions to complete the trial
5. Patients who signed an informed consent form.

Healthy Subjects:

1. No abnormalities on cranial
2. 18-80 years old
3. Able to complete cognitive task
4. Able to follow instructions to complete the trial
5. not taking medications.
6. Subjects who signed an informed consent form.

Exclusion Criteria:

Stroke patients:

1. Inability to tolerate the test due to organic diseases
2. Serious mental illness that prevents them from cooperating with or tolerating the trial
3. Pregnant or lactating women
4. Had metal implants, a history of other neurological disorders, acute cardiopulmonary dysfunction.

Healthy Subjects:

1. Inability to tolerate the test due to organic diseases
2. Serious mental illness that prevents them from cooperating with or tolerating the trial.
3. Pregnant or lactating women
4. Had metal implants, a history of other neurological disorders, acute cardiopulmonary dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with stroke in the inpatient ward of the Department of Rehabilitation Medicine, The First Affiliated Hospital of Chongqing Medical University.
  Healthy subjects recruited through the Department of Rehabilitation Medicine, The First Affiliated Hospital of Chongqing Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Preliminary screening of brain function biomarkers for post-stroke cognitive impairment | 1 day
  Comparison of differences in brain activation [HbO2 (mmol/L*mm)] between patients with post-stroke cognitive impairment and patients without post-stroke cognitive impairment or healthy subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Medicine, the First Affiliated Hospital of Chongqing Medical University, Chongqing,, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided